CLINICAL TRIAL: NCT03679819
Title: Single-center Trial for the Validation of High-resolution Transrectal Ultrasound (Exact Imaging Scanner ExactVu) for the Detection of Prostate Cancer
Acronym: EXACTVU
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Institut Paoli-Calmettes (Other)
Collaborators: Exact Imaging (Industry)
Responsible Party: Sponsor
Other Study IDs: EXACTVU-IPC 2016-019; 2017-A01745-48 (Other: ANSM IDRCB)
Record Dates: First submitted 2018-09-17; First posted 2018-09-20 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Prostate Cancer
Keywords: multiparametric MRI; ExactVu ultrasound scanner; prostatectomy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HR-TRUS: HR-TRUS for the detection of prostate cancer in men scheduled for radical prostatectomy for localized prostate cancer
  Interventions: Device: HR-TRUS

INTERVENTIONS:
Device: HR-TRUS — Medical procedures to be performed in the study consist of subject preparation and prostate imaging. The HR-TRUS exam will be done with a transrectal probe either the day before surgery, or in the OR right before surgery. The exam will be done in the same manner as during a regular transrectal ultrasound exam and no invasive procedures will be associated.

SUMMARY:
The primary objective of this study is to evaluate the performance of HR-TRUS in detection of prostate cancer lesions relative to whole mount section after radical prostatectomy as the reference.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the performance of HR-TRUS in detection of prostate cancer lesions relative to whole mount section after radical prostatectomy as the reference. The analysis will include the detection of all prostate cancer lesions as well as the detection of significant prostate cancer lesions. With this approach it is possible to calculate the sensitivity, specificity, negative predictive value, positive predictive value and overall accuracy of the correct detection of prostate cancer in the prostate. These results are of importance when the ExactVu ultrasound scanner is to be used later for prostate cancer diagnosis using targeted biopsies.

ELIGIBILITY:
Inclusion Criteria:

1. men > 35 years age and <80 years of age
2. diagnosed with prostate cancer by prostate biopsy scheduled for radical prostatectomy
3. staging by standard procedures show localized disease (<cT4)
4. PSA < 50ng/ml
5. Access to the rectum for trans rectal ultrasound
6. Patient affiliated to the ''National security'' regimen or beneficiary of this regimen
7. Signed written informed consent prior to any screening procedures being performed

Exclusion Criteria:

1. Patient with absence of diagnosis of prostate cancer
2. Patient with metastatic prostate cancer
3. Patient with rectal amputation
4. Patient with contraindications for MRI
5. Patient in urgency situation, adult under legal protection, or unable to give his consent.

Ages: 35 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — male patients that are diagnosed with localized prostate cancer
Study Population: The study population will consist of male patients that are diagnosed with localized prostate cancer by prostate biopsy and that are scheduled for radical prostatectomy as treatment for their disease.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-09-05 (Actual); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of high resolution ultrasound | From date of HR-TRUS exam until the date of Prostate biopsy data are obtained (average of 7 days)
  rate of adequately identified (positive or negative) lesions of prostate cancer

SECONDARY OUTCOMES:
Precisions of high-resolution ultrasound and multiparametric MRI in the detection of lesions of prostate cancer. | From date of HR-TRUS exam until the date of Prostate biopsy data are obtained (average of 7 days)
  sensitivity, specificity, negative and positive predictive values of high-resolution ultrasound and multiparametric MRI in the detection of lesions of prostate cancer.
Morphology of lesions not detected by high-resolution ultrasound | From date of HR-TRUS exam until the date of Prostate biopsy data are obtained (average of 7 days)
  Volume and grade of lesions not detected by high-resolution ultrasound
Localization of lesions not detected by high-resolution ultrasound | From date of HR-TRUS exam until the date of Prostate biopsy data are obtained (average of 7 days)
  Location of lesions not detected by high-resolution ultrasound
Extra-prostatic extensions detected by high-resolution ultra-sound | From date of HR-TRUS exam until the date of Prostate biopsy data are obtained (average of 7 days)
  Extra-prostatic extensions and seminal vesicle invasions detected by high-resolution ultra-sound in positive and negative sectors

CONTACTS AND LOCATIONS:
Overall Officials: Jochen Walz, MD, Principal Investigator — Institut Paoli-Calmettes
Locations (1):
- Institut Paoli Calmettes, Marseille, Bouches Du Rhone, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pavlovich CP, Cornish TC, Mullins JK, Fradin J, Mettee LZ, Connor JT, Reese AC, Askin FB, Luck R, Epstein JI, Burke HB. High-resolution transrectal ultrasound: pilot study of a novel technique for imaging clinically localized prostate cancer. Urol Oncol. 2014 Jan;32(1):34.e27-32. doi: 10.1016/j.urolonc.2013.01.006. Epub 2013 Apr 2. PMID 23558161
- [Background] Walz J, Marcy M, Maubon T, Brunelle S, Laroche J, Gravis G, Salem N, Bladou F. [Real time elastography in the diagnosis of prostate cancer: comparison of preoperative imaging and histology after radical prostatectomy]. Prog Urol. 2011 Dec;21(13):925-31. doi: 10.1016/j.purol.2011.04.006. Epub 2011 Jun 2. French. PMID 22118357
- [Background] Ghai S, Eure G, Fradet V, Hyndman ME, McGrath T, Wodlinger B, Pavlovich CP. Assessing Cancer Risk on Novel 29 MHz Micro-Ultrasound Images of the Prostate: Creation of the Micro-Ultrasound Protocol for Prostate Risk Identification. J Urol. 2016 Aug;196(2):562-9. doi: 10.1016/j.juro.2015.12.093. Epub 2016 Jan 12. PMID 26791931
- [Background] Boehm K, Salomon G, Beyer B, Schiffmann J, Simonis K, Graefen M, Budaeus L. Shear wave elastography for localization of prostate cancer lesions and assessment of elasticity thresholds: implications for targeted biopsies and active surveillance protocols. J Urol. 2015 Mar;193(3):794-800. doi: 10.1016/j.juro.2014.09.100. Epub 2014 Sep 28. PMID 25264337
- [Background] Villers A, Puech P, Mouton D, Leroy X, Ballereau C, Lemaitre L. Dynamic contrast enhanced, pelvic phased array magnetic resonance imaging of localized prostate cancer for predicting tumor volume: correlation with radical prostatectomy findings. J Urol. 2006 Dec;176(6 Pt 1):2432-7. doi: 10.1016/j.juro.2006.08.007. PMID 17085122